CLINICAL TRIAL: NCT00964132
Title: A Multiple-Center, Open-Label, Study of the Safety and Efficacy of Oral NRX 194204 Capsule Administered Daily for a Minimum of 4 Weeks in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Oral NRX 194204 Study in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NuRx Pharmaceuticals, Inc. (Industry)
Responsible Party: Roshantha A. Chandraratna, PhD, MBA, Chief Scientific Officer, NuRx Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 194204-203
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Rexinoid; NRX194204; Lung Cancer; RXR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — AGN 194204

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NRX194204 (Experimental)
  Interventions: Drug: NRX194204

INTERVENTIONS:
Drug: NRX194204 — Once Daily, Oral

SUMMARY:
The purpose of this study is to determine whether NRX 194204 is effective in the treatment of advanced Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Numerous studies in pre-clinical models and in human clinical trials have clearly established the potential for the use of rexinoids in the treatment and prevention of cancer. NRX 194204, a second generation rexinoid, is a highly potent and specific activator of RXRs. Because NRX 194204 is significantly more selective for the RXRs relative to the RARs than a first generation approved drug, it is associated with fewer adverse events in clinical use. This study seeks to investigate NRX 194204 monotherapy in patients who have failed any 2 prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years
* Histologically confirmed advanced stage III or IV NSCLC that is recurrent or has progressed after treatment. Failure on at least 2 NSCLC treatment regimens
* Uni-dimensionally measurable NSCLC defined as at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as ≥ 2cm with conventional techniques or as ≥ 1cm on spiral CT scan.
* Patients are eligible if disease free from previous malignancies, other than a previous NSCLC, for greater than two years. Patients with a history of prior basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix are not excluded.
* Karnofsky performance status ≥ 60 (Attachment 14.4) or ECOG performance status 0-2
* Life expectancy > 12 weeks.
* Able to swallow capsule form of the drug.
* Hematology:

  * Hemoglobin > 8.5 g/dl;
  * Platelets > 100,000 cells/mm3;
  * Neutrophils > 1500 cells/mm3;
  * PT and PTT within normal limits, except for patients receiving Coumadin for thromboembolic prophylaxis only, in whom INR of less than 2 will be allowable.
* Biochemistry:

  * Total bilirubin < 1.5 x ULN;
  * AST/ALT < 3.0 x ULN;
  * Serum creatinine < 2.0 mg/dl;
  * Serum calcium < 11.5 mg/dl;
  * Fasting serum triglycerides < 2.5 x ULN.
* Negative urine pregnancy test for women of child-bearing potential at screening and on Day 1, and agreement by both women and men of reproductive potential to use two reliable forms of contraception during therapy and for 1 month following discontinuation of therapy unless abstinence is the chosen birth control method.
* Able to follow study instructions, accessible for treatment and follow-up, and likely to complete all study requirements.

Exclusion Criteria:

* Significant medical history or unstable medical condition (congestive heart failure, recent myocardial infarction within 3 months, unstable angina, active systemic infection, uncontrolled hypertension). Patients with controlled diabetes will be allowed.
* Prior treatment with bexarotene (Targretin) or NRX 194204.
* Current enrollment in an investigational drug or device study or participation in such a study within 21 days of entry into this study.
* Known sensitivity to any of the ingredients in the study medication.
* Known HIV-positive patients.
* Females who are pregnant, nursing, or planning a pregnancy.
* Major surgery within previous 4 weeks; large field radiation therapy (> 25% of the patient's total marrow) or chemotherapy (including investigational agents or participation in another clinical study) within previous 3 weeks; mitomycin C or nitrosoureas within 6 weeks. In all instances, patients must have fully recovered from acute toxicities related to prior therapies.
* Systemic retinoid therapy, or Vitamin A at dosages > 15,000 IU per day, during previous 4 weeks.
* Patients with a history of pancreatitis or at significant risk of developing pancreatitis (e.g., uncontrolled hyperlipidemia, excessive alcohol consumption, uncontrolled diabetes mellitus, and medications known to increase triglyceride levels or to be associated with pancreatic toxicity).
* Primary brain tumors, active brain metastasis including progression from last scan or evidence of cerebral edema, or clinical symptoms of brain metastasis.
* Condition or situation which, in the investigator's opinion, may put patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Overall objective tumor response rate | 7 months

SECONDARY OUTCOMES:
Progression free survival | 7 months
Overall survival | 7 months
Overall safety and toxicity of NRX 194204 in NSCLC patients | 7 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Dr. Pandit, Fountain Valley, California
  - UCSD Moores Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Somerset Oncology Hematology Associates, Somerville, New Jersey
  - Swedish Cancer Institute, Seattle, Washington